CLINICAL TRIAL: NCT05491941
Title: Assessment for Implementation Methods in Sepsis
Acronym: AIMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Levy, Director of Critical Care Medicine at Lifespan, and Chief of the Division of Pulmonary, Critical Care and Sleep Medicine, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HL162954-01 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Sepsis Severe; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Hybrid 2 implementation effectiveness trial with a cluster randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hour-1 Bundle (Active Comparator): If the patient meets 2+ SIRS and chief complaint criteria, a second BPA may be triggered, which displays to the provider. The second alert identifies patients who progress to organ failure based on lab results, or who have a recorded instance of hypotension. When this alert appears, an automatic counter will begin and serve as our Sepsis Time Zero. The provider will receive sepsis order sets and guided to the Sepsis Navigator. The navigator will allow them to review relevant patient data, reference sepsis guidelines, and keep tabs on a live-updating sepsis checklist to ensure they complete each element in order and on time. Following identification in the ED, both study arms will receive the same bundle (see below). The only difference will be the timing: For the Hour-1 bundle, all interventions in the bundle must be initiated within 1 hour.
  Interventions: Other: Sepsis Bundle
- 3-Hour Bundle (Active Comparator): If the patient meets 2+ SIRS and chief complaint criteria, a second BPA may be triggered, which displays to the provider. The second alert identifies patients who progress to organ failure based on lab results, or who have a recorded instance of hypotension. When this alert appears, an automatic counter will begin and serve as our Sepsis Time Zero. The provider will receive sepsis order sets and guided to the Sepsis Navigator. The navigator will allow them to review relevant patient data, reference sepsis guidelines, and keep tabs on a live-updating sepsis checklist to ensure they complete each element in order and on time. Following identification in the ED, both study arms will receive the same bundle (see below). The only difference will be the timing: For the 3-hour bundle, all elements must be completed by 3 hours.
  Interventions: Other: Sepsis Bundle

INTERVENTIONS:
Other: Sepsis Bundle — Intervention initiated within 1 hour or 3 hours of presentation depending on the Arm: 1. Measure lactate level. 2. Obtain blood cultures before administering antibiotics. 3. Administer broad-spectrum antibiotics. 4. Begin rapid administration of 30ml/kg crystalloid for hypotension or lactate greater than or equal to 4mmol/L. 5. Apply vasopressor if hypotensive during or after fluid resuscitation to maintain a mean arterial pressure greater than or equal to 65 mm Hg.

SUMMARY:
Since the introduction of sepsis bundles, there have been multiple published trials that have demonstrated a consistent, strong association between implementation of sepsis "bundles" (3-hour bundle) and improved survival. The current proposal is a Hybrid 2, pragmatic, cluster randomized clinical effectiveness/implementation trial evaluating mortality and respiratory failure-based outcomes, in patients admitted to the emergency department with sepsis, comparing the effectiveness of implementation of the hour-1 bundle to 3-hour bundle, while facilitating adherence to both bundles. In addition, 4 distinct sepsis phenotypes will be derived from routine clinical data to identify specific patient phenotypes that allow for a more precision-based application of sepsis bundles in future studies.

DETAILED DESCRIPTION:
Sepsis is the leading cause of admission to intensive care units (ICUs) in the U.S., and the leading cause of respiratory failure and death in ICUs. The majority of ICU patients with sepsis or septic shock have either respiratory infection as the source of sepsis, or have respiratory failure requiring mechanical ventilation. In recognition of the burden of sepsis in the U.S., sepsis "bundles" were introduced to facilitate guideline implementation in clinical practice (known as the 3-Hour bundle). Since the introduction of sepsis bundles, multiple observational studies have demonstrated a consistent, strong association between implementation of sepsis bundles and improved survival. These data led to the New York State (NYS) Sepsis initiative, which demonstrated a significant association between adherence with sepsis bundles and improved survival, and the Centers for Medicare and Medicaid Services (CMS) mandated public reporting of sepsis measures (SEP-1). Analysis of the NYS database has revealed that completion of the 3-Hour bundle in patients with respiratory failure was associated with an 8.6% absolute reduction in mortality (18.5 RRR). For those patients who completed the 3-Hour bundle within 1 hour, the mortality reduction was even higher, 9.8% (RRR 21.7%). In 2018, the Hour-1 bundle was published to underscore the need for urgency in the treatment of septic patients. We believe that the primary beneficial effect of both the Hour-1 and 3-Hour bundle is in patients with respiratory failure. It is not known if implementation of the Hour-1 bundle reduces mortality more than the 3 Hour bundle. Although adherence with the 3-Hour bundle (SEP-1) is mandated by CMS, compliance is moderate (60%), suggesting an active implementation process for the 3-hour bundle is necessary to compare the Hour-1 bundle to the 3-Hour bundle. The current proposal is a pragmatic, cluster-randomized clinical trial using a hybrid type 2 effectiveness-implementation approach to evaluate mortality and respiratory failure-based outcomes and bundle adherence, in emergency room patients with sepsis. We will compare the hour-1 bundle to the 3-hour bundle. The outcome measures include hospital mortality, hospital length of stay, ventilator-free days, and incidence of respiratory failure. The effectiveness of a clinical intervention (Hour-1 bundle) is implemented using a rigorous implementation strategy (the Exploration, adoption/Preparation, Implementation, Sustainment - EPIS - multi-level conceptual model) for both the 1- and 3-Hour bundles. We will also evaluate a possible precision-based approach in this study. Routine clinical information available at hospital presentation will identify 4 discrete, sepsis phenotypes and we hypothesize that 2 of these identify patients who are significantly more likely to benefit from the 1-Hour bundle in future studies. Our team has extensive experience conducting multi-center trials in sepsis guided by effective models of implementation science. We have developed automated screening tools to identify patients with sepsis and have guided state-wide implementation of sepsis performance measures. We have also used automated EHR methods to screen for and enroll septic patients into these studies. This novel, hybrid type 2 effectiveness-implementation approach addresses key gaps to facilitate the implementation of evidence-based strategies to improve patient outcomes from sepsis and acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18
* Patient meets criteria for time zero (sepsis within 6 hours of ED triage and the 3 criteria-infection, 2 SIRS and 1 or more organ dysfunctions, must be met within 3 hours of each other.

Exclusion Criteria:

* Last admission for patients admitted to same hospital once
* Pregnant women
* All transfers from another hospital
* Individuals who are made comfort care only within 6 hours of admission to ED
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  Mortality associated with death from sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Levy, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frank HE, Evans L, Phillips G, Dellinger R, Goldstein J, Harmon L, Portelli D, Sarani N, Schorr C, Terry KM, Townsend SR, Levy MM. Assessment of implementation methods in sepsis: study protocol for a cluster-randomized hybrid type 2 trial. Trials. 2023 Sep 29;24(1):620. doi: 10.1186/s13063-023-07644-y. PMID 37773067